CLINICAL TRIAL: NCT05479110
Title: The Effectiveness of Using Empathy Experience Courses to Guide Occupational Therapy Students in Case-base Clinical Reasoning- A Pilot Study
Brief Title: The Effectiveness of Using Empathy Courses to Guide OT Students in Case-base Clinical Reasoning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMU-JIRB N202112011
Record Dates: First submitted 2022-06-21; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-06

CONDITIONS: Students

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group was given four 3-hour training sessions over 2 weeks, which included group instruction on empathy experience, clinical reasoning, and functional therapy case-oriented learning.
  Interventions: Behavioral: Empathy experience courses and case-base clinical reasoning
- Control group (Active Comparator): The control group was given case studies(text).
  Interventions: Other: case studies

INTERVENTIONS:
Behavioral: Empathy experience courses and case-base clinical reasoning — Four 3-hour training sessions over 2 weeks, which included group instruction on empathy experience, clinical reasoning, and functional therapy case-oriented learning.
  Arms: Experimental group
Other: case studies — active control: case studies(text)
  Arms: Control group

SUMMARY:
Clinical reasoning is an important cognitive process in medical decision making. In recent years, medical education advocates holistic medicine, but systematic learning is rare in school education.Therefore, this study used an empathy experience course to conduct a case-oriented clinical reasoning training course to improve the empathy and clinical reasoning skills of pre-clinical students in occupational therapy through four sessions.

DETAILED DESCRIPTION:
Objective: To investigate effectiveness of using empathy experience courses to guide the students who prior to occupational therapy(OT) practice in case-base clinical reasoning.

Materials and Methods: 30 students were recruited from 8 universities in Taiwan and randomly divided into an experimental group and a control group. The experimental group was given four 3-hour training sessions over 2 weeks, which included group instruction on empathy experience, clinical reasoning, and functional therapy case-oriented learning, while the control group was given case studies. Tests were administered before and after the series of sessions, including case report writing, C-JES-HPS, SACRR, and a follow-up visit at the end of the first phase of clinical practice using the C-JES-HPS and SACRR; course satisfaction surveys were completed after each session and at the follow-up visit to observe course satisfaction, usefulness, and recommendations. Data were analyzed using SPSS (version 20.0) with a significance level of 0.05. Univariate analyses with repeated measures 2-way analysis of variance were used to compare changes in empathy and clinical reasoning ability between the two groups of subjects and course satisfaction was presented as descriptive statistics. It was hypothesized that a case-oriented clinical reasoning training program using an empathy experience program would improve empathy and clinical reasoning skills in pre-practicum students in occupational therapy.

ELIGIBILITY:
Inclusion Criteria:

* Occupational therapy students from National Taiwan University, Kaohsiung Medical University, Sun Yat-sen Medical University, National Cheng Kung University, Chang Gung University, IShou University, Fu Jen Catholic University, and Asia University who have completed their major credits and will be interning in a clinical hospital.
* Must be at least 20 years old and under 65 years old.

Exclusion Criteria:

* Those who are unable to attend the whole course.
* Those who have not completed their school credits and are unable to go to the clinical hospital for internship.
* Those who do not speak Chinese or English as their native language.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Chinese version of the Jefferson Scale of Empathy-Health Profession Students | Change from Baseline at 2 weeks
  A total of 20 questions were used to self-assess participants' empathy status and were scored using a 7-point Likert scale. The content covered three sections, including 10 questions on the perspective taking section, 8 questions on the compassionate care section, and 2 questions on standing in the patient's shoes.
The Self-Assessment of Clinical Reflection and Reasoning | Change from Baseline at 2 weeks
  A 26-item, five-point Likert scale was used to self-assess clinical reasoning skills, including strongly disagree, disagree, unsure, agree, and strongly agree.

SECONDARY OUTCOMES:
Satisfaction Questionnaire | up to 2 weeks
  The researchers designed the form to understand the subjects' satisfaction with the content of the training course, the usefulness of the training course for clinical practice, and their suggestions for the training course. Satisfaction with the content of the training course and the usefulness of the training course for clinical practice were rated on a five-point Likert scale of very dissatisfied, dissatisfied, fair, satisfied, and very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Hanyun Hsiao, Principal Investigator — Taipei Medical University, Taiwan, R.O.C.
Locations (1):
- Taipei Medical University Shuang Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Addy TM, Hafler J, Galerneau F. Faculty Development for Fostering Clinical Reasoning Skills in Early Medical Students Using a Modified Bayesian Approach. Teach Learn Med. 2016 Oct-Dec;28(4):415-423. doi: 10.1080/10401334.2016.1186551. Epub 2016 Jun 9. PMID 27283028
- [Background] Cooper N, Bartlett M, Gay S, Hammond A, Lillicrap M, Matthan J, Singh M; UK Clinical Reasoning in Medical Education (CReME) consensus statement group. Consensus statement on the content of clinical reasoning curricula in undergraduate medical education. Med Teach. 2021 Feb;43(2):152-159. doi: 10.1080/0142159X.2020.1842343. Epub 2020 Nov 18. PMID 33205693
- [Background] Daniel M, Rencic J, Durning SJ, Holmboe E, Santen SA, Lang V, Ratcliffe T, Gordon D, Heist B, Lubarsky S, Estrada CA, Ballard T, Artino AR Jr, Sergio Da Silva A, Cleary T, Stojan J, Gruppen LD. Clinical Reasoning Assessment Methods: A Scoping Review and Practical Guidance. Acad Med. 2019 Jun;94(6):902-912. doi: 10.1097/ACM.0000000000002618. PMID 30720527
- [Background] Duca NS, Glod S. Bridging the Gap Between the Classroom and the Clerkship: A Clinical Reasoning Curriculum for Third-Year Medical Students. MedEdPORTAL. 2019 Jan 25;15:10800. doi: 10.15766/mep_2374-8265.10800. PMID 31139730
- [Background] Huhn K, Gilliland SJ, Black LL, Wainwright SF, Christensen N. Clinical Reasoning in Physical Therapy: A Concept Analysis. Phys Ther. 2019 Apr 1;99(4):440-456. doi: 10.1093/ptj/pzy148. PMID 30496522
- [Background] Jamieson M, Krupa T, O'Riordan A, O'Connor D, Paterson M, Ball C, Wilcox S. Developing empathy as a foundation of client-centred practice: evaluation of a university curriculum initiative. Can J Occup Ther. 2006 Apr;73(2):76-85. doi: 10.2182/cjot.05.0008. PMID 16680911
- [Background] Min Simpkins AA, Koch B, Spear-Ellinwood K, St John P. A developmental assessment of clinical reasoning in preclinical medical education. Med Educ Online. 2019 Dec;24(1):1591257. doi: 10.1080/10872981.2019.1591257. PMID 30935299
- [Background] Posel N, Mcgee JB, Fleiszer DM. Twelve tips to support the development of clinical reasoning skills using virtual patient cases. Med Teach. 2015;37(9):813-8. doi: 10.3109/0142159X.2014.993951. Epub 2014 Dec 19. PMID 25523009
- [Background] Svalastog AL, Donev D, Jahren Kristoffersen N, Gajovic S. Concepts and definitions of health and health-related values in the knowledge landscapes of the digital society. Croat Med J. 2017 Dec 31;58(6):431-435. doi: 10.3325/cmj.2017.58.431. No abstract available. PMID 29308835
- [Background] Ten Cate O. Competency-Based Postgraduate Medical Education: Past, Present and Future. GMS J Med Educ. 2017 Nov 15;34(5):Doc69. doi: 10.3205/zma001146. eCollection 2017. PMID 29226237
- [Background] Wenham J, Best M, Kissane DW. Systematic review of medical education on spirituality. Intern Med J. 2021 Nov;51(11):1781-1790. doi: 10.1111/imj.15421. PMID 34142417